CLINICAL TRIAL: NCT02403713
Title: A Randomised, Open-label, 2-group PK (3-period) and PD (5-period) Crossover Study to Compare Systemic Exposure and Pharmacodynamic Effects of Fluticasone/Formoterol BAI and pMDI in Healthy Volunteers
Brief Title: A Pharmacokinetic/Pharmacodynamic Inhaler Comparison Study in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mundipharma Research Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KFL1503; 2013-000045-39 (EudraCT Number)
Record Dates: First submitted 2015-02-19; First posted 2015-03-31 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Fluticasone; Formoterol Fumarate; Metered Dose Inhalers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Test Treatment (Experimental): Fluticasone/formoterol 125/5 µg BAI
  Interventions: Drug: Fluticasone/formoterol BAI
- Active Comparator 1 (Active Comparator): Fluticasone/formoterol 125/5 µg pMDI with spacer
  Interventions: Drug: Fluticasone/formoterol PMDI with spacer
- Active Comparator 2 (Active Comparator): Fluticasone/formoterol 125/5 µg pMDI without spacer
  Interventions: Drug: Fluticasone/formoterol PMDI without spacer
- Active Comparator 3 (Active Comparator): Fluticasone/formoterol pMDI (125/5 μg) without spacer, low dose
  Interventions: Drug: Fluticasone/formoterol PMDI without spacer low dose
- Active Comparator 4 (Active Comparator): Formoterol (12 µg) without spacer
  Interventions: Drug: Formoterol

INTERVENTIONS:
Drug: Fluticasone/formoterol BAI — Fluticasone/formoterol 125/5 µg breath actuated inhaler (BAI) (250/10 µg total dose)
  Arms: Test Treatment
Drug: Formoterol — Formoterol
  Arms: Active Comparator 4
Drug: Fluticasone/formoterol PMDI without spacer — Fluticasone/Formoteral 125/5µg pMDI without spacer
  Arms: Active Comparator 2
Drug: Fluticasone/formoterol PMDI with spacer — Fluticasone/Formoteral 125/5µg pMDI with spacer
  Arms: Active Comparator 1
Drug: Fluticasone/formoterol PMDI without spacer low dose — Fluticasone/Formoteral 125/5µg pMDI without spacer, low dose
  Arms: Active Comparator 3

SUMMARY:
A 2-group healthy volunteer study to compare a breath actuated inhaler (BAI) and a pressurised metered dose inhaler (pMDI) with and without spacer.

DETAILED DESCRIPTION:
Group 1 will assess pharmacokinetics, Group 2 will assess pharmacodynamics. PK interim analysis to determine requirement for PK extension.

Group 1 (PK) blood sampling and safety assessments up to 36 hours post-dose for 3 study periods. Results from PK stage will determine if Group 2 (PD) is required. Group 2 (PD) will assess LABA only effects (as confirmed in interim analysis).

Group 2 (PD) to include 2 overnight stays for 5 study periods. Volunteers will receive a single dose of study medication, with discharge on Day 2.

Study treatments are fluticasone/formoterol BAI, fluticasone/formoterol pMDI with/without spacer, formoterol alone without spacer, and low dose fluticasone/formoterol without spacer.

Volunteers will undergo blood sampling, and safety assessments up to the morning of discharge. An inspiratory flow recorder (IPR) will be used for training and to monitor inspiratory flow rate, inhaled volume and inhalation technique.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18 years or over.
* Healthy and free of significant abnormal findings as determined by medical history, physical examination, vital signs, laboratory tests and ECG.
* Normal lung function (FEV1 >90% of predicted normal value).
* Demonstrate satisfactory technique in the use of the study drug devices.
* No use of steroid medication (systemic or topical) within 8 weeks prior to study screening.

Exclusion Criteria:

* Subjects who use any asthma medication or are knowingly regularly exposed to asthma medication.
* Any history of drug or alcohol abuse.
* Any history of conditions that might interfere with drug absorption, distribution, metabolism or excretion.
* History of asthma, COPD, or other bronchial or lung diseases.
* User of steroid medication (systemic or topical) within 8 weeks prior to study screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2014-08; Primary Completion 2014-10 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters Composite measurement of Pharmacokinetic parameters (Cmax, AUCt, AUCINF). | Pre dose to 36 hours post dose
Serum Potassium | Pre Dose to 6 hours post first dose
  Maximum reduction in serum potassium from pre-dose.

SECONDARY OUTCOMES:
Vital Signs | Pre Dose to 6 hours post dose
  Composite measurement of vital signs (heart rate and blood pressure)
Serum Glucose | Pre Dose to 6 hours post dose
  Maximum increase in Serum Glucose

CONTACTS AND LOCATIONS:
Locations (1):
- Belfast, United Kingdom